CLINICAL TRIAL: NCT04902664
Title: A Multi-pronged Intervention to Initiate Shared Decision-making on Medical Tests and Care Cascades in the Primary Care Setting
Brief Title: Shared Decision-making on Medical Tests and Care Cascades
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: RAND (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Ishani Ganguli MD, MPH, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P001080
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Health Knowledge, Attitudes, Practice; Health Care Utilization
MeSH Terms: conditions — Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: 20 primary care physicians will be recruited and randomized to an intervention and a control arm. For each physician, we will recruit at least 10 of their patients with upcoming scheduled physicals. All included patients of intervention physicians will receive the intervention, and all included patients of control physicians will receive general patient visit prep materials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Intervention arm physicians will receive an email with feedback on how they compare to their peers in aggregate on test ordering during annual physicals, along with physician-facing education materials. This email will be sent before each patient study visit for all patients in the study. Participating patients of intervention arm physicians will receive patient education materials one to two days before their study visit.
  Interventions: Behavioral: Patient education materials; Behavioral: Physician peer-comparison email; Behavioral: Physician education materials
- Control Arm (Placebo Comparator): Control arm physicians receive an email with information on the general visit preparation tips that their patients will receive. Participating patients of control arm physicians will receive general visit preparation tips one to two days before their study visit.
  Interventions: Behavioral: General visit preparation materials

INTERVENTIONS:
Behavioral: Patient education materials — Patients receive a text-message and email with educational materials about medical testing.
  Arms: Intervention Arm
Behavioral: Physician peer-comparison email — Physicians receive an email with feedback on how they compare to their peers in aggregate on test ordering during annual physicals.
  Arms: Intervention Arm
Behavioral: Physician education materials — Physicians receive reference materials on medical test interpretation and incidental findings.
  Arms: Intervention Arm
Behavioral: General visit preparation materials — Patients receive a text-message and email with general visit preparation tips.
  Arms: Control Arm

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the impact of patient and provider facing educational materials and peer comparison on medical testing conversations during annual physicals. The investigators hypothesize that education materials and peer comparison will improve conversation quality about medical testing decisions.

DETAILED DESCRIPTION:
Medical tests may show unexpected findings leading to additional tests, treatments, and visits that cost money and take time but may not have benefits. This is a prevalent issue with major consequences for patients and clinicians. Making informed decisions about when to order medical tests may help avoid unnecessary costs and worry. However, doctors don't always have detailed conversations about medical testing and there are patient gaps in knowledge. The investigators hypothesize that education materials and peer comparison to promote conversations about medical tests will improve conversation quality about medical testing decisions. The investigators have developed patient and provider-facing interventions to educate on and promote conversations about the uses and consequences of medical tests, and the investigators will test the impact of this just-in-time educational and peer comparison intervention on the likelihood of patients having productive conversations about medical tests. The effects of the intervention will be assessed using surveys before and after the study. This work has the potential to help patients feel more supported by their healthcare system, empower patients to participate in shared decision-making, and build trust between patients and clinicians.

ELIGIBILITY:
Inclusion criteria (Physicians):

* Primary care physicians at Brigham and Women's Hospital
* In active practice

Inclusion criteria (Patients):

* Adults age 18 years old or older
* English-speaking
* Access to email
* Did not opt out of receiving research invitations from health system
* Patients of participating physicians
* Scheduled annual physical during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Shared Decision-Making Process 4 Survey | Within two weeks after visit
  Composite score of survey items completed by the patient after physician visit. Min 0, Max 4 (higher is better).

SECONDARY OUTCOMES:
Presence of testing discussion | Within two weeks after visit
  Binary measure from patient post-visit survey (present vs absent)
Satisfaction with testing discussion | Within two weeks after visit
  Binary measure from patient post-visit survey (high vs low)
Discussion of next steps | Within two weeks after visit
  Binary measure from patient post-visit survey (present vs absent)
Whether doctor explained tests in a way that was easy to understand | Within two weeks after visit
  Binary measure from patient post-visit survey (yes completely vs yes a little or no)
Patient knowledge | Within two weeks after visit
  Composite score of survey items from patient post-visit survey. Min 0, Max 4 (higher is better).

CONTACTS AND LOCATIONS:
Overall Officials: Ishani Ganguli, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Robert S Rudin, PhD, Principal Investigator — RAND
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganguli I, Mulligan KL, Chant ED, Lipsitz S, Simmons L, Sepucha K, Rudin RS. Effect of a Peer Comparison and Educational Intervention on Medical Test Conversation Quality: A Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2342464. doi: 10.1001/jamanetworkopen.2023.42464. PMID 37943557